CLINICAL TRIAL: NCT01473654
Title: Avoiding Diabetes Thru Action Plan Targeting (ADAPT): A Pilot Randomized Control Trial of an Electronic Medical Record Embedded Prediabetes Shared Goal Setting Tool in Primary Care
Brief Title: The Avoiding Diabetes Thru Action Plan Targeting Pilot Randomized Control Trial
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-30397; 5K23DK081665 (NIH)
Record Dates: First submitted 2011-11-15; First posted 2011-11-17 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADAPT tool (Experimental): prediabetes counseling using ADAPT tool
  Interventions: Behavioral: ADAPT tool
- Control (No Intervention)

INTERVENTIONS:
Behavioral: ADAPT tool — Use of ADAPT shared goal setting tool in EMR
  Other Names: ADAPT
  Arms: ADAPT tool

SUMMARY:
The goal of this randomized control trial is to study the impact of an electronic health record embedded tool's ability to facilitate shared provider-patient goal setting to promote lifestyle behavior change and prevent diabetes in primary care.

DETAILED DESCRIPTION:
The ADAPT (Avoiding Diabetes Thru Action Plan Targeting) trial is an innovative study that leverages persuasive technology to enhance the lifestyle behavior change counseling efficacy of primary care providers. Using principles of behavior change theory and persuasion technology, the multidisciplinary design team utilized in-depth interviews and in-vivo usability testing to produce a prototype diabetes prevention counseling system embedded in the electronic health record. The core element of the tool is a streamlined shared goal setting module within the electronic health record system. The system also utilizes a pre-encounter patient behavior change goals elicitation survey to help tailor the goal setting session to patient preferences and encourage shared decision making. The patients also interact with a website that collects their longitudinal behavior change data and visualizes their progress over time and in comparison to other study members. The ADAPT system utilizes the influential powers of goal setting, tailoring, reminders, social comparisons, testimonials and other methods to integrate evidence based behavior change principles and persuasion techniques into routine primary care clinical encounters. If successful, the ADAPT system may represent an adaptable and scalable technology-enabled behavior change tool for all primary care providers.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes

Exclusion Criteria:

* age<18
* diabetes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 6 months
  measured by pedometer

SECONDARY OUTCOMES:
hemoglobin a1c | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Devin Mann, MD, MS, Principal Investigator — Boston University
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Mann DM, Lin JJ. Increasing efficacy of primary care-based counseling for diabetes prevention: rationale and design of the ADAPT (Avoiding Diabetes Thru Action Plan Targeting) trial. Implement Sci. 2012 Jan 23;7:6. doi: 10.1186/1748-5908-7-6. PMID 22269066